CLINICAL TRIAL: NCT04507438
Title: The Effect of Donepezil on Glycemic Control in Type II Diabetics
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen Wills, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH201804
Record Dates: First submitted 2020-03-05; First posted 2020-08-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Donepezil; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Donepezil treatment group (Experimental): Administration of 5mg or 10 mg of donepezil daily
  Interventions: Drug: Donepezil 5-10 Mg Oral Tablet
- Control group (Placebo Comparator): Administration of placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Donepezil 5-10 Mg Oral Tablet — Donepezil 5mg or 10mg oral tablet administered daily for an 8 week period
  Arms: Donepezil treatment group
Drug: Placebo Oral Tablet — Placebo oral tablet administered daily for an 8 week period
  Arms: Control group

SUMMARY:
The purpose of the study is to establish the effectiveness of the drug Donepezil in treating Type 2 Diabetes Mellitus compared to a control treatment. Donepezil is not approved by the FDA to treat Type 2 Diabetes Mellitus and its use in this research is experimental. 50 patients with Type 2 Diabetes Mellitus (Adult Onset Diabetes Mellitus) will be randomized to either the donepezil treatment group or the control group after screening. (25 patients in each arm; a total of 50 patients). Both men and women shall be enrolled.Donepezil shall be orally administered to the study group. Control group will get an orally administered placebo which is an inert compound, lactose. Wk0 will be the randomization visit. The patients will take the drug for 8 weeks and the last follow up visit will be the last day of week 8.

DETAILED DESCRIPTION:
The study is a randomized, double blinded, treatment-controlled, parallel design to investigate the effect of donepezil (administration of 5-10 mg of donepezil daily, orally, over 8 week period) on clinical outcomes reflecting diabetic control. The research assistant will not be blinded. The investigator and patient shall be blinded. A computer program will be used to randomize the patients.

50 patients with Type 2 Diabetes Mellitus (Adult Onset Diabetes Mellitus) will be randomized to either the donepezil treatment group or the control group after screening. (25 patients in each arm; a total of 50 patients). Both men and women shall be enrolled.

As many patients as required to meet the enrollment numbers shall be screened. Patients will be monitored daily for blood pressure, glucose levels and heart rate, during the period of hospitalization. Adjustments in insulin or oral hypoglycemic, blood pressure and heart rate control medications will occur during this time. Follow up visits will be made as required and at the end of week 8.

Donepezil shall be orally administered to the study group. Control group will get an orally administered placebo which is an inert compound, lactose.

Wk0 will be the randomization visit. The patients will take the drug for 8 weeks and the last follow up visit will be the last day of week 8.

Any anticholinergic drugs will be eliminated from the patients' medical regimen with the exception for inhaled anticholinergic. There is no known major contraindication of acetylcholinesterase inhibitors (like for eg: galantamine, rivastigmine and donepezil) Patients shall be monitored closely for vagotonic effect. Acetylcholine is known to have a vagotonic effect lowering heart rate and blood pressure. Therefore, during the course of administration of the drug close attention to heart rate and blood pressure will be a significant part off the clinical management of patients. If the patients are on beta blockers, their beta blocker dose will be closely monitored and adjusted as required.

Proton pump inhibitors will be used to guard against any possible GI bleed. 40 mg of pantoprazole once daily.

Patient will be observed for seizures. The patients will be examined for pulmonary exacerbation during treatment in the hospital. If the pulmonary status deteriorates they will be eliminated from the study. The medication administration will not start sooner than 24 hrs after surgery. Patients shall be observed for exaggerated response from anesthesia.

Only lipid profile and fasting blood sugar has to be done fasting. As many tests as possible shall be combined and done at the same time to avoid multiple needle pricks to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 50 with Type 2 Diabetes Mellitus, regardless of co-morbidities including renal and vascular insufficiency, Cardiovascular Autonomic Neuropathy, Hypertension, Chronic Obstructive Pulmonary Disease or Coronary Disease will be selected.

Exclusion Criteria:

* Patients under the age of 50
* Patients who are pregnant or lactating
* Patients who are lactose intolerance
* Patients with an allergy to Donepezil
* Prothrombin Time and International Normalized Ratio value greater than 1.25
* Pre-menopausal women and patients allergic to Donepezil are excluded.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C | 8 weeks

SECONDARY OUTCOMES:
Change in blood urea nitrogen | 8 Weeks
  Change will be assessed by reviewing blood urea nitrogen/creatinine
Change in creatinine | 8 weeks
  Change will be assessed by reviewing blood urea nitrogen/creatinine

OTHER OUTCOMES:
Change in lipid profile | 8 Weeks
Change in albumin | 8 weeks
  Weight and albumin will be monitored to asses change in nutritional status

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Shore Regional Health, Easton, Maryland, United States